CLINICAL TRIAL: NCT06616727
Title: A Phase I Study to Evaluate the Safety, Tolerability and Pharmacokinetics of SNC109 in Patients With Recurrent Glioblastoma
Brief Title: The Safety and Efficacy of SNC-109 CAR-T Cells Therapy the rGBM
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Simnova Biotechnology Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNC109-102
Record Dates: First submitted 2024-09-02; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Recurrent Glioblastoma Multiforme (GBM)
Keywords: GBM
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SNC109 CART (Experimental): After the screening and evaluation, SNC-109 CAR-T Cells will be infusion.
  Interventions: Drug: SNC109

INTERVENTIONS:
Drug: SNC109 — SNC-109 CAR-T Cells, first dose from 5×104 CAR+ T Cells, treatment follows the operation and the next dose would be deiced by SRC

SUMMARY:
A phase I study to evaluate the safety, tolerance and pharmacokinetics of SNC109 in patients with rGBM

DETAILED DESCRIPTION:
It is planned to recruit about 50 patients with rGBM subjects. The protocol consists of screening period, Lymphocytes apheresis period, Operation period, pre-infusion evaluation (-2~-1 days), infusion (day 0), infusion observation (day 1-post infusion), and follow-up period (last infusion-720 days). The incidence of dose limitation toxicity (DLT) will be observed within 28 days after the first infusion. Subjects in this study will receive multiple infusions, starting with 5×104 CAR+ T cells/dose in the first subject, and the Safety Review Committee (SRC) will evaluate the subsequent dosing regimen, dose, infusion interval, and number of treatment cycles. Subsequent subjects will be evaluated by the SRC on the basis of available PK and safety data, and the SRC will determine the dosing regimen, dose, infusion interval and number of treatment cycles based on observed evidences.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18，both sexes;
* Diagnosed with a history of glioblastoma, and the recurrent glioblastoma has confirmed by histological/molecular pathology (including astrocytoma World Health Organization (WHO) Grade 4);
* Karnofsky (KPS) ≥50;
* The estimated survival time is ≥12 weeks;
* Blood pregnancy tests for women of childbearing age are negative;
* The patient himself/herself, and/or his/her legal guardian, agree to participate in the trial and sign the informed consent form.

Exclusion Criteria:

* Known allergies to study drugs or drugs that may be used in the study;
* Severe concurrent diseases in the heart, lungs, liver, or other vital organs;
* Hypertension is poorly controlled or accompanied by hypertensive crisis or hypertensive encephalopathy;
* In addition to the glioblastoma, with other severe central nervous system diseases or complications or aggressive malignancies;
* Long-term use of immunosuppressant drugs, or large doses of steroids;
* Received live or attenuated vaccine or other surgery had no related to GBM within 4 weeks prior to Lymphocytes apheresis;
* Lymphocytes apheresis or cell infusion combined with infection or unexplained fever.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-26 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment related adverse events | Up to 28 days after first infusion
  Incidence of adverse events associated with CAR-T cell transfusion within 28 days of the first infusion, abnormal and clinical significant laboratory results
DLT | Up to 28 days after first infusion
  Incidence of DLT associated with CAR-T cell transfusion within 28 days of the first infusion

SECONDARY OUTCOMES:
Overall survival (OS) after infusion | within 2 years after first infusion
  The data of Overall survival (OS) after infusion
Time maximum of SNC-109 Cell count and CAR vector copy number | within 2 years after first infusion
  Pharmacokinetic (PK) profile/parameter Tmax
Pharmacokinetic (PK) profile/parameters Peak Plasma Concentration (Cmax) of SNC-109 Cell count and CAR vector copy number | within 2 years after first infusion
  Peak Plasma Concentration (Cmax)
Pharmacokinetic (PK) profile/parameters Area under the plasma concentration versus time curve (AUC) | within 2 years after first infusion
  Area under the plasma concentration versus time curve (AUC) of SNC-109 Cell count
Progression free survival (PFS) after infusion | within 2 years after first infusion
  The data of Overall survival (OS) after infusion
Efficacy assesment for the treatment according to iRANO | within 2 years after first infusion
  Assessment of disease response rates according to the Immunological Response Assessment in Neuro-Oncology (iRANO)
Pharmacodynamic (PD) profile/parameters Changes of Cytokines after infusion | within 2 years after first infusion
  Changes of cytokines (such as Interleukin-6, Interleukin-8 etc.) in peripheral blood (PB) and cerebrospinal fluid (CSF) pre-and post- infusion and at each of the main follow-up time points, and the time to recovery
Concentration of Human anti-chimeric antibody (HACA) | within 2 years after first infusion
  Detection of changes in peripheral blood and cerebrospinal fluid Human anti-chimeric antibody (HACA)

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, China